CLINICAL TRIAL: NCT07074210
Title: Value of Volume Oxygenation Index to Detect Early Failure of Non-invasive Ventilation in Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Entsar Hsanen, Principal investigator, Assiut University
Other Study IDs: volume oxygenation index COPD
Record Dates: First submitted 2025-06-28; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: COPD; Non Invasive Ventilation (NIV); VOX Index
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: non invasive ventilation — Non invasive mechanical ventilation pressure support

SUMMARY:
Non-invasive ventilation (NIV) is an evidence-based treatment for patients with acute respiratory failure due to an exacerbation of Chronic Obstructive Pulmonary Disease (COPD). In patients with COPD and acute hypercapnic respiratory failure, NIV improves gas exchange, reduces the work of breathing, and decreases the length of hospital stay and mortality [1]. Furthermore, when compared to invasive ventilation, NIV leads to fewer complications, such as ventilator-related infections [2]. These findings have resulted in guideline recommendations for the use of NIV in acute respiratory failure due to an exacerbation of COPD [3].NIV failure has been defined as the need for endotracheal intubation (ETI) or death. Its rate varies greatly between 5% and 60%, depending on numerous factors [4].

The Volume Oxygenation (VOX) index, initially developed to predict treatment failure of high flow nasal cannula therapy, has demonstrated the ability to estimate early increases in respiratory drive. Within the first 2 h, the VOX index exhibits a discriminative potential of 0.88 (95 % CI 0.79-0.97) in predicting HFNC failure [5]. Based on this premise, we hypothesize that the VOX index could be a predictive tool for NIV treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with COPD admitted to the respiratory ICU for NIV.

Exclusion Criteria:

* Patients indicated for urgent intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be subjected to Complete history taking, including demographic characteristics, diagnosis on admission to the hospital, length of ICU stay, length of hospital stay, and chronic underlying diseases. Vital signs, complete lab investigation, APACHE II, and SOFA score will be collected. Non-invasive pressure support ventilation (PSV) mode will be used, using pressure support 15 mmH2o to calculate the VTm (average of three consecutive VT monitoring values / Predicted Body Weight). Arterial blood gases will be collected at admission, and within 2 hours of NIV, and after 24h of NIV to calculate the VOX index [6].
  VOX index =SpO2 / (FiO2 * VTm).
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Need for Invasive mechanical ventilation | 1 week
  deterioration and invasive ventilation

SECONDARY OUTCOMES:
in hospital mortality | 1 week
  patient death

IPD SHARING:
Plan to Share IPD: Undecided